CLINICAL TRIAL: NCT04846374
Title: Two is Better Than One: A Novel Venous Access System for Intermittent Apheresis
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: 21-0287
Record Dates: First submitted 2021-04-13; First posted 2021-04-15 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Apheresis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- PowerPort Subjects: This study will involve a chart review of patients at UNC who were referred for change from a vortex port to a powerflow port.
  Interventions: Device: PowerPort

INTERVENTIONS:
Device: PowerPort — The study will compare pheresis sessions with the old system versus pheresis sessions with one of two new configurations.

SUMMARY:
Purpose: To describe a novel configuration of venous access for the performance of intermittent apheresis.

Participants: 20 participants at UNC who were referred for change from a vortex port to a powerflow port.

Procedures (methods): Placement of one of two configurations of the powerflow port and follow up visits between January 1, 2019 and December 31, 2023.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18 years of age.
* Referred for change from a vortex port to a powerflow port.
* Previously placed or scheduled placement of one of two configurations of the PowerFlow port

Exclusion Criteria:

* Unable to read and understand English.
* Unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 20 adults will be enrolled to this study. The study subjects will be recruited from adults who are scheduled to receive or have received a PowerFlow™ Implantable Apheresis IV Port in Vascular Interventional Radiology for their clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-04-14 (Actual)

PRIMARY OUTCOMES:
Change in Flow Rate | 1 year following new port configuration placement
  The study will compare mean change flow rate for pheresis sessions with the old system versus pheresis sessions with one of two new configurations by averaging the flow rate for up to 5 sessions using the new port configuration.
Change in Procedure Time | 1 year following new port configuration placement
  The study will compare mean change in procedure time for pheresis sessions with the old system versus pheresis sessions with one of two new configurations.

SECONDARY OUTCOMES:
Change in Use of Tissue Plasminogen Activator | 1 year following new port configuration placement
  The study will compare mean change in use of tissue plasminogen activator for pheresis sessions with the old system versus pheresis sessions with one of two new configurations.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bream, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol
Time Frame: 9 to 36 months following publication
Access Criteria: The investigator who proposes to use the data has received IRB, IEC, or REB approval, as applicable, and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Derived] Howlett MS, Hicks K, Park Y, Karafin MS, Bream PR Jr. Use of a novel configuration of ports for patients needing intermittent long-term apheresis. J Clin Apher. 2024 Aug;39(4):e22143. doi: 10.1002/jca.22143. PMID 39105402